CLINICAL TRIAL: NCT07201038
Title: Feasibility of Ultrafast WGS in Paediatric Malignancies
Brief Title: Ultrafast Whole Genome Sequencing for Childhood Cancer
Acronym: UF-WGS
Status: Recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Illumina, Inc. (Industry); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Aditi Vedi, Chief Investigator, University of Cambridge
Other Study IDs: IRAS317008
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cancer Childhood
Keywords: whole genome sequencing
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — extracted DNA will be stored
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrafast WGS cohort, prospective patients
- Ultrafast WGS, retrospective patients

SUMMARY:
Cambridge University Hospitals NHS Foundation Trust (CUHNFT) is the Principal Treatment Centre for the East of England region, responsible for 120-150 patients <16 years with a new diagnosis of paediatric malignancy annually; leukaemia comprises ~25% of these cases. Current molecular diagnosis of subgroups of childhood malignancies, particularly leukaemia, is based on flow cytometry, fluorescent in situ hybridisation (FISH) and single nucleotide polymorphim (SNP) arrays, for which the usual turnaround time (TAT) is 7-14 days. In the current era of access to targeted therapy, rapid diagnosis and treatment of patients in high-risk molecular subgroups is critical for improving outcomes. Children and adolescents with Philadelphia-chromosome positive (Ph+) acute lymphoblastic leukaemia (ALL) have significantly improved survival when treated with tyrosine kinase inhibitors (TKIs). Patients with Ph+-like mutations (10- 20% of paediatric ALL), also have a poor prognosis, requiring escalation of treatment and addition of targeted therapy. Rapidly identifying MYCN amplification is also of critical prognostic importance in embryonal tumours of childhood including neuroblastoma (25%) and medulloblastoma, and directly impacts on treatment from the outset of the patient journey. Overnight whole genome sequencing (WGS) entails taking an additional 5ml Peripheral Blood (PB) and Bone Marrow (BM) samples after samples for routine diagnostic workup have been collected, and could replace current standard of care (SOC), which has a median turnaround time (TAT) of up to 28 days, and up to 84 days for specific gene mutations, which can delay appropriate prognostication and management of high-risk patients. Rapid, point of care information on somatic and germline mutations will allow early risk stratification and expedite treatment for high-risk patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate
* Be aged <25 years of age
* Have confirmed or suspected malignancy
* For pilot/feasibility study (first 10 patients), only haematological malignancies (ALL/AML) will be included
* Have tumour and germline sample available - retrospectively collected or for prospective collection

Exclusion Criteria:

* Inability to provide written informed consent (self or parent/guardian)
* Insufficient tissue (BM/PB/tissue) available for research purposes after collection for routine diagnostic purposes

Ages: 0 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with cancer at relapse or initial diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2027-10-18 (Estimated); Study Completion 2028-10-17 (Estimated)

PRIMARY OUTCOMES:
turnaround time from sample collection to availability of meaningful results. | 36 months

SECONDARY OUTCOMES:
Percentage of enrolled patients with available WGS results from the Ultrafast WGS pipeline. | 24 months
Correlation of data from Ultrafast WGS against current SOC WGS data. | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided